CLINICAL TRIAL: NCT06427837
Title: Child Snack Variety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutritional Sciences, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ChildFood802
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Same 2nd course (Experimental): The same snack food will be served in the second course
  Interventions: Other: Same 2nd course
- Different 2nd course (Experimental): A different snack food will be served in the second course
  Interventions: Other: Different 2nd course

INTERVENTIONS:
Other: Same 2nd course — The same snack food will be served in the second course
  Arms: Same 2nd course
Other: Different 2nd course — A different snack food will be served in the second course
  Arms: Different 2nd course

SUMMARY:
The purpose of this study is to determine how consumption of a snack food at a first course affects the hedonic ratings of that snack food compared to other foods, and how it affects intake of a second course. The results will have implications for guidance about the provision of snacks for preschool children and may help in identifying strategies for the prevention of obesity in children.

ELIGIBILITY:
Inclusion Criteria:

* Children who are enrolled in a participating childcare center
* Children who are between the ages of 6 and 14 years old at the time of enrollment

Exclusion Criteria:

* Children who are allergic to any of the foods served
* Children whose diets exclude any of the foods served
* Children who are absent from the childcare center on study days
* Children who are not able to complete study measures (e.g. refuse to eat study foods, only use the anchors or have low variability for their liking ratings, etc.)

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Change between interventions of snack intake by weight | Study weeks 1 and 2
  Weight (grams) of food and water consumed
Change between interventions of snack intake by energy | Study weeks 1 and 2
  Energy (kcal) of food consumed

SECONDARY OUTCOMES:
Change between interventions in liking of each test food | Study weeks 1 and 2
  Change between interventions in liking (before to after consumption) of the 5 test foods, measured using a visual analog scale (0-100 points).
Change between interventions in ranked preference of each test food from before to after consumption | Study weeks 1 and 2
  Change in ranked preference (before to after consumption) of the 5 test foods.
Change between interventions in fullness ratings from before to after consumption | Study weeks 1 and 2
  Change in fullness ratings (before to after consumption) measured using a 4-point scale ranging from empty to full.

CONTACTS AND LOCATIONS:
Locations (1):
- 311 Chandlee Laboratory, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No